CLINICAL TRIAL: NCT06978920
Title: A Phase I, Open Label, Single Arm, Dose Escalation and Dose Expansion Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Human Induced Pluripotent Stem Cell Derived Dopaminergic Progenitor Cells (NCR201) Injection in the Treatment of Subjects With Parkinson's Disease
Brief Title: A Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of NCR201 in the Treatment of Subjects With Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCR201-2001
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose (Experimental): MRI-guided bilateral stereotactic cell implantation
  Interventions: Drug: Allogeneic dopaminergic neural precursor cell(NCR201)
- High Dose (Experimental): MRI-guided bilateral stereotactic cell implantation
  Interventions: Drug: Allogeneic dopaminergic neural precursor cell(NCR201)

INTERVENTIONS:
Drug: Allogeneic dopaminergic neural precursor cell(NCR201) — Bilateral implantation

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and preliminary efficacy that NCR201 has on Parkinson's disease (PD) patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disease in the middle-aged and elderly. It is the "third killer" of the middle-aged and elderly after tumors and cardiovascular and cerebrovascular diseases. Its main clinical manifestations are resting tremor, reduced voluntary movement, muscle rigidity, postural reflex impairment, and autonomic dysfunction, which seriously affect patients' work ability and quality of life. It is estimated that nearly 100,000 people in China become new Parkinson's patients every year. Experts from the World Health Organization predict that the number of Parkinson's patients in China will reach 5 million in 2030, which will be more than half of the world's total. As the disease progresses, the symptoms of Parkinson's patients will become increasingly severe. The high prevalence and high disability rate of Parkinson's disease bring heavy burdens to individuals, families, and society.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 40 and 75 years;
* Diagnosed to be Parkinson's disease according to Parkinson's disease diagnostic criteria;
* Disease history over 5 years;
* Stable dose of dopamine treatment;
* Able to undergo PET/CT/MRI detection;

Exclusion Criteria:

* Patients who have previously undergone brain surgery;
* Past use of stem cell therapy or participation in stem cell clinical research;
* Cognitive impairment;
* History of mental disorders;
* Patients with other serious systemic diseases;
* Past or current metastatic malignant tumors.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | Within 24 weeks post-transplantation
  Safety and tolerability

SECONDARY OUTCOMES:
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part III, in comparison with baseline values. | Within 24 months post-transplantation
  Minimum score: 0; Maximum score: 132; Higher scores mean a worse outcome.
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part I,II,IV, in comparison with baseline values. | Within 24 months post-transplantation
  Higher scores mean a worse outcome.
Assessment of changes in Hoehn & Yahr scale in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in Parkinson disease.
Assessment of changes in Hamilton Depression Scale (HAMD)-17 in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in mental state.
Assessment of changes in Hamilton Anxiety Scale (HAMA)-14 in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in mental state.
Assessment of changes in Parkinson's Disease Questionnaire-39 (PDQ-39) in comparison with baseline values. | Within 24 months post-transplantation
  Comprehensive clinical assessment for examining the improvements in activity of daily living.
Bilateral putamen standardized uptake value as demonstrated on positron emission tomography(PET) compared with baseline in the 'off' state. | Within 24 months post-transplantation
  Evidence of cell survival
Patient L-dopa equivalent dose compared with baseline. | Within 24 months post-transplantation
  Measure of dopaminergic drug dose
Incidence and severity of adverse events. | Within 24 months post-transplantation
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No